CLINICAL TRIAL: NCT01596127
Title: Safety and Efficacy of Intrathecal Rituximab in Patients With Lymphoid Malignancies Involving the Central Nervous System
Brief Title: Intrathecal Rituximab in Lymphoid Malignancies Involving Central Nervous System
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0844; NCI-2012-00849 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Leukemia; Lymphoid Malignancies; Metastatic Malignant Neoplasm to the Leptomeninges
Keywords: relapsed CD20+ lymphoid malignancies; refractory CD20+ lymphoid malignancies; Rituximab; Intrathecal Rituximab; CNS; Leptomeningeal disease; LMD; central nervous system disease; Relapsed lymphoid malignancies; refractory lymphoid malignancies; CNS leukemia; intrathecal chemotherapy; cerebrospinal fluid; CSF; lumbar puncture; LP
MeSH Terms: conditions — Leukemia; Meningeal Carcinomatosis; Meningeal Neoplasms; Central Nervous System Diseases | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intrathecal Rituximab (Experimental): Phase I Starting Dose: Rituximab administered via lumbar puncture at dose of 10 - 25 mg twice weekly according to the dose escalation.
  Phase II Rituximab Starting Dose: Maximum tolerated dose from Phase I.
  Interventions: Drug: Intrathecal Rituximab

INTERVENTIONS:
Drug: Intrathecal Rituximab — Phase I: Starting dose Rituximab 10 mg intrathecally twice weekly until 2 consecutive CSF samples are negative for the presence of blast cells. Thereafter, rituximab 10 mg intrathecally weekly for additional 4 weeks, followed by intrathecal rituximab 10 mg administered once every other week for an additional 8 weeks.
  Phase II Starting Dose of Rituximab: Maximum tolerated dose from Phase I.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn about the safety and effectiveness of rituximab given by spinal tap in patients with lymphoid malignancies involving the central nervous system.

A spinal tap (also called a lumbar puncture) is when fluid surrounding the spinal cord is collected by inserting a needle into the lower back. The affected area is numbed with local anesthetic during the procedure. It will also be used to give chemotherapy in this study.

Rituximab is designed to bind to a protein, called CD20, that is on the surface of the leukemia cells. This may cause the leukemia cells to die.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

If you are found to be eligible, you will be assigned to a study group based on when you join this study. Up to 12 participants will be enrolled in the Phase I portion of the study, and up to 13 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of rituximab you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of rituximab. Each new group will receive a higher dose of rituximab than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of rituximab is found.

If you are enrolled in the Phase II portion, you will receive rituximab at the highest dose that was tolerated in the Phase I portion.

Study Visits:

Once enrolled, you will return to the clinic and receive the study drug by spinal tap up to 2 times a week. You will receive treatment twice a week until 2 CSF samples in a row do not show any leukemia cells. After that, you will receive treatment 1 time a week for an additional 4 weeks, and then you will receive treatment once every other week for an additional 8 weeks. The number of doses you receive will depend on how many doses the study doctor thinks is needed.

At each study visit the following procedures will be performed:

* You will have a physical exam, including measurement of your weight, and vital signs. °Your vital signs will be measured every 15 minutes for 1 hour after each dose of rituximab.
* You will be asked how well you are able to perform the normal activities of daily living (performance status).
* You will be asked about any drugs you may be taking and any side effects you may experiencing.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* A sample of cerebral spinal fluid may be collected from the lumbar puncture to verify the absence or presence of blast cells.

Follow-Up:

About 30 days after your last dose of study drug you will be contacted by the study staff by telephone and asked about any drugs you may be taking and any side effects you may experiencing. This call should take about 10 minutes.

Long-term Follow-up:

Every 6 to 12 months you may be contacted by the study staff by telephone and asked about any drugs you may be taking and any side effects you may experiencing. This call should take about 10 minutes.

You may be given other drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Length of Treatment:

The number of treatments you receive will depend on how long it takes for there to be no leukemia cells in the CSF samples. Once this happens, you will have treatments for an additional 12 weeks. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Rituximab is FDA approved and commercially available for the treatment of relapsed and/or refractory lymphoid malignancies involving the central nervous system. Receiving rituximab by spinal tap is considered investigational.

Up to 25 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have relapsed or refractory CD20+ lymphoid malignancies with either documented CNS involvement or peripheral nerve infiltration.
2. Patients 3 years of age and older are eligible after 3 patients (age 15 or older) have been treated and did not experience a dose limiting toxicity. Patient 3 to 15 years of age will follow the dose escalation schema independent of the adults.
3. ECOG performance status measure will be used. (ECOG Performance Status less than or equal to 3)
4. Adequate liver function (bilirubin less than or equal to 3 mg/dL within 24 hours of enrollment)
5. Adequate renal function (serum creatinine less than or equal to 3 mg/dL within 24 hours of enrollment)
6. Urine pregnancy test for women of childbearing potential (defined as not post-menopausal for 12 consecutive months or no previous surgical sterilizations). A negative urine pregnancy test is required within 48 hours of initiating study drug.
7. Signed informed consent

Exclusion Criteria:

1. Known active meningeal infection
2. History of severe infusion reaction to any monoclonal antibody

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: 1/24/2013 through 11/13/2013. All participants recruited at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Four patients were enrolled and three participants were evaluable for safety and efficacy and toxicity. One patient was ineligible and therefore was never treated. Due to lack of response and slow accrual, the study was terminated early.
Groups:
- Intrathecal Rituximab: Phase I Starting Dose: Rituximab administered via lumbar puncture at dose of 10 - 25 mg twice weekly according to the dose escalation.
  Phase II Rituximab Starting Dose: Maximum tolerated dose from Phase I.
  Intrathecal Rituximab: Phase I: Starting dose Rituximab 10 mg intrathecally twice weekly until 2 consecutive CSF samples are negative for the presence of blast cells. Thereafter, rituximab 10 mg intrathecally weekly for additional 4 weeks, followed by intrathecal rituximab 10 mg administered once every other week for an additional 8 weeks.
  Phase II Starting Dose of Rituximab: Maximum tolerated dose from Phase I.
Period: Overall Study
Arm/Group | Intrathecal Rituximab
Started | 4
Completed | 3
Not Completed | 1
Not completed — Patient Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intrathecal Rituximab
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 38 [31 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The percentage of participants whose cancer shrinks or disappears after treatment where participants are considered as responding to therapy if the Cerebrospinal fluid (CSF) is without evidence of blast cells after four lumbar punctures with rituximab.
Time Frame: 2 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | Intrathecal Rituximab
Number analyzed (Participants) | 3
percentage of Participants | 0

2. Secondary Outcome: Maximum Tolerated Dose (MTD) of Rituximab
Description: MTD is dose level at which at least 1 of 3 participants experiences a dose-limiting toxicity (DLT). DLTdefined as clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and meeting the NCI common terminology criteria that are CTCAE Grade 3 or 4.
Time Frame: 2 weeks
Population: Multiple dose levels were designed with a starting dose of 10 mg per injection followed by 25 mg once safety was established in the first 3 patients treated at the first dose level. The study moved tot he next dose level. Due to lack of response and slow accrual, participants were never treated on the next dose level and the study was terminated
Arm/Group | Intrathecal Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug.
Arm/Group | Intrathecal Rituximab
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Rituximab (N=3)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Multi-organ Failure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Rituximab (N=3)
Spasticity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Headache (General disorders) | 3 (3)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-04-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT01596127/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT01596127/SAP_001.pdf